CLINICAL TRIAL: NCT04402151
Title: Single-Arm Phase II Study of PSMA PET/MR Guided Stereotactic Body Radiation Therapy With Simultaneous Integrated Boost (SBRT-SIB) for High-Intermediate and High Risk Prostate Cancer
Brief Title: Study of PSMA PET/MR Guided Stereotactic Body Radiation Therapy With Simultaneous Integrated Boost (SBRT-SIB) for High-Intermediate and High Risk Prostate Cancer
Acronym: PSMA SBRT-SIB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Telix Pharmaceuticals (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-10020928; R01CA249615 (NIH)
Record Dates: First submitted 2020-05-08; First posted 2020-05-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Other): Patients enrolling on the protocol will undergo prostate-specific membrane antigen (PSMA) Positron Emission Tomography (PET)/Magnetic Resonance(MR) prior to start of the radiation treatment planning process. PSMA tracer is administered by IV injection and PET images are acquired.
  Any patients found to have possible metastatic disease will undergo a standard of care confirmatory biopsy (if feasible) and receive treatment appropriate for their stage.
  The PSMA PET/MR scan will be performed prior to initiation of androgen deprivation therapy (ADT).
  Interventions: Drug: PSMA PET/MR - Gallium-68 labeled PSMA-HBED-CC; Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: PSMA PET/MR - Gallium-68 labeled PSMA-HBED-CC — Patients enrolling on the protocol will undergo prostate-specific membrane antigen (PSMA) Positron Emission Tomography (PET)/Magnetic Resonance(MR) prior to start of the radiation treatment planning process. PSMA tracer is administered by IV injection and PET images are acquired.
  Any patients found to have possible metastatic disease will undergo a standard of care confirmatory biopsy (if feasible) and receive treatment appropriate for their stage.
  The PSMA PET/MR scan will be performed prior to initiation of androgen deprivation therapy (ADT).
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Patients will receive standard of care radiation therapy (SBRT)

SUMMARY:
This is a single-arm Phase II clinical trial assessing the clinical efficacy of prostate specific membrane antigen (PSMA) PET/MR guided MR-LINAC based SBRT-SIB with planned accrual of 50 patients.

DETAILED DESCRIPTION:
Localized prostate cancer can be treated in 5 sessions using a precise, targeted form of radiation known as stereotactic body radiation therapy (SBRT), with low toxicity. Despite these advances, overall outcomes for aggressive (high risk) prostate cancer remain poor, with 10-year recurrence-free survival of approximately 65% regardless of treatment modality. Recurrences are typically distant and carry poor prognosis, with 5 year survival of 25%. The investigators propose to utilize the latest advances in cancer imaging (PSMA Positron Emission Tomography (PET)/Magnetic Resonance Imaging (MR)) and radiation delivery (MR-guided radiation therapy with real-time adaptive planning), to deliver a personalized radiation treatment that targets the areas of greatest risk of recurrence in the prostate with improved precision, and as a result improve clinical outcomes for individuals with high risk prostate cancer. PSMA PET/MR is a novel imaging modality, not yet widely available, that augments the tissue detail provided by MR. The combination of PSMA PET with MR results in improved delineation of intraprostatic nodules and higher diagnostic accuracy for detection of metastatic disease compared to conventional imaging. PSMA PET/MR imaging data is readily transferable to a MR-based linear accelerator (MR-LINAC), a novel, innovative platform that allows direct visualization of the tumor during treatment, and permits real-time individualized correction for motion with online adaptive radiation planning.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 21 years or older.
* Ability to provide signed informed consent and willingness to comply with protocol requirements.
* Pathologic confirmation of high-risk adenocarcinoma of the prostate gland as follows: a. Gleason 8-10 or tertiary component 5 disease and/or b. PSA of 20 ng/ml or greater and/or c. Tumor stage of T2c or greater; OR Unfavorable intermediate risk (Gleason 4+3=7, >50% of cores involved, or 2 or more intermediate risk factors which include Gleason 7 disease, PSA 10-20, or T2b disease)
* Participants must agree to use an acceptable form of birth control and utilize condoms for a period of seven days after each PSMA injection, if engaged in sexual activity.
* No evidence of metastatic disease, including pelvic lymph nodes.

Exclusion Criteria:

* Clinical and/or technical factors that would compromise statistical analysis of the PET and/or MR.
* Contraindications to PSMA IV administration
* Contraindications to prostate SBRT (history of transurethral resection of prostate; prostate size greater than 150 cc; AUA score greater than 20; history of prior radiation to the prostate)
* Other unspecified reasons that, in the opinion of investigators, make the subject unsuitable for enrollment
* Patients on or intending to take abiraterone will be excluded

Ages: 21 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients
Enrollment: 50 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy of prostate-specific membrane antigen (PSMA) Positron Emission Tomography (PET)/Magnetic Resonance(MR), MR-Linear Accelerator (LINAC) will be assessed by evaluating recurrence free survival | 24 months
  Evaluate the clinical efficacy of PSMA PET/MR guided, MR-LINAC-based SBRT- SIB in high-intermediate and high risk prostate cancer, as evaluated by the 2-year recurrence-free survival rate

SECONDARY OUTCOMES:
Performance of PSMA PET/MR to MR alone at staging prostate cancer | Baseline
  Detection of metastatic disease on each scan will be recorded, with pathologic confirmation obtained. Detection of intraprostatic nodules will be recorded with pathologic confirmation obtained.
Performance of PSMA PET/MR to MR alone for identification of dominant intraprostatic nodules during radiation planning | Baseline
  The Dominant Intraprostatic Nodules (DIN) will be defined with radiologist assistance on MR alone, and subsequently PSMA PET/MR. The incidence of alterations in target will be recorded.
Compare imaging biomarkers of interest on MR and PSMA PET/MR as predictors of treatment response, versus biopsy of treatment response and PSA | Baseline
Compare imaging biomarkers of interest on MR and PSMA PET/MR as predictors of treatment response, versus biopsy of treatment response and PSA | 12 months
Change in Quality of life questionnaires (EPIC-26) will be assessed. | Baseline, 1month, 6months, 12 months, 18 months and 24 months.
  Expanded Prostate Cancer Index Composite (EPIC) short form questionnaire. The Expanded Prostate Cancer Index Composite (EPIC) is a comprehensive instrument designed to evaluate patient function and bother after prostate cancer treatment. Scores range from 0 to 100, lower scores indicate worse outcomes and higher EPIC scores represent better outcomes.
Change in The American Urological Association (AUA) symptom score | Baseline, 1month, 6months, 12 months, 18 months and 24 months.
  The American Urological Association (AUA) has created this symptom index for understanding the severity of enlarged prostate symptoms. Scores ranging from 0-7 are considered to be mild symptoms, 8-19 are moderate and 20 - 35 are severe symptoms.
Change in Number of Subjects with Adverse events | Baseline, 1month, 6months, 12 months and 24 months.
  Adverse events will be collected from patients based on CTCAE version 5.0.
The change in radiation doses received by the surrounding normal structures/PTV for each initial and adapted plan will be analyzed with a signed-rank Wilcoxon test (non-parametric test for paired comparisons). | Baseline, 1month
  PTV is the planning target volume
Compare the changes in the Microbiome during SBRT-SIB | Baseline
  Gut microbiome samples will be obtained for 16S RNA analyses
Compare the changes in the Microbiome during SBRT-SIB | approx. 3 weeks
  Gut microbiome samples will be obtained for 16S RNA analyses
Compare the changes in the Microbiome during SBRT-SIB | 12 months
  Gut microbiome samples will be obtained for 16S RNA analyses
Compare the immunological changes during SBRT-SIB | Baseline
  serum samples will be obtained for immune correlate analyses
Compare the immunological changes during SBRT-SIB | approx. 3 weeks
  serum samples will be obtained for immune correlate analyses
Compare the immunological changes during SBRT-SIB | 12 months
  serum samples will be obtained for immune correlate analyses

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Formenti, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No